CLINICAL TRIAL: NCT05904574
Title: Evaluation of the the Effectiveness of the Autologous Blood Patch Method in Transthoracic Lung Biopsies Using the Coaxial Technique
Brief Title: Effectiveness of the Autologous Blood Patch Method in Lung Biopsies
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burak USLU, Principal investigator, Trakya University
Other Study IDs: TTLBABPTU21
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; Pneumothorax
Keywords: lung cancer; pneumothorax; computed tomography; biopsy
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: The patients who underwent tru-cut biopsy with the coaxial technique and applied an autologous blood patch.
  Interventions: Other: Autologous blood patch; Other: Percutaneous transthoracic biopsy
- B: The patients whose true-cut biopsy with coaxial technique was taken and autologous blood patch was not applied.
  Interventions: Other: Percutaneous transthoracic biopsy

INTERVENTIONS:
Other: Autologous blood patch — Approximately 3-4 pieces were taken with the 18 G core biopsy needle until sufficient tissue was obtained. In the autologous blood patch technique, approximately 6-7 ml of blood was taken from the patient with a 10 ml syringe before the procedure. By attaching a 3-way tap to the injector from which the blood is drawn, blood is drawn into a second injector to ensure that the clotted blood is dispersed and homogenized. The prepared autologous blood patch was given through the coaxial needle (approximately 1 ml of autologous blood patch was applied for every 1 cm when the coaxial needle was withdrawn) and the tract formed by the biopsy needle in the parenchyma, pleura, and under the skin was closed with the patient's autologous blood.
  Groups: A
Other: Percutaneous transthoracic biopsy — After determining the lung lobe where the lesion was observed, axial CT images of 5 mm cross-section thickness were obtained so that the upper and lower parts of it could be visualized. After ruling the entry site in the skin, antisepsis and local anesthesia were performed. The coaxial system (17 G) was cautiously advanced and CT images were continuously evaluated to confirm entrance into the lesion. Biopsy was taken and after sufficient tissue samples were taken at the last stage of the biopsy procedure, control CT imaging, including the whole lung, was performed to evaluate complications. The presences of pneumothorax were noted.

SUMMARY:
In this retrospective study, investigators aimed to evaluate the effectiveness of the autologous blood patch method in percutaneous transthoracic lung biopsies performed with the coaxial technique.

DETAILED DESCRIPTION:
In this retrospective study, investigators aimed to evaluate the effectiveness of the autologous blood patch method in percutaneous transthoracic lung biopsies performed with the coaxial technique. Biopsies and treatment modalities were performed according to approved guidelines. Ethics committee approval was obtained for the retrospective evaluation of the files and images of the participants. Written informed consent was obtained from all participants before biopsy procedures. Percutaneous transthoracic biopsies (PTB) have been started to be performed with the coaxial technique using the autologous blood patch method as of April 2019 in Interventional Radiology Department of Trakya University Hospital. All lung biopsies are performed using the blood patch method as a standard, as a clear decrease in procedural complications was observed in a short time. Thus, in this study, participants who underwent biopsy after April 2019 formed the participant group that underwent autologous blood patch, and those who had the procedure before this date formed the control group. Since autologous blood patch application was not performed before this date, participant grouping was time-dependent.

All participants included in the study underwent tru-cut biopsy with the coaxial technique. Of the 240 participants included in the study, 120 were treated with an autologous blood patch ( Group A), and the remaining 120 were participants without an autologous blood patch (Group B).

Procedure:

All biopsy procedures were performed by four interventional radiologists with at least 2 years of experience. First of all, after determining the lung lobe where the lesion was observed, axial CT images of 5 mm cross-section thickness were obtained so that the upper and lower parts of it could be visualized. After ruling the entry site in the skin, antisepsis and local anesthesia were performed. The coaxial system (17 G) was cautiously advanced and CT images were continuously evaluated to confirm entrance into the lesion. Approximately 3-4 pieces were taken with the 18 G core biopsy needle until sufficient tissue was obtained. In the autologous blood patch technique, approximately 6-7 ml of blood was taken from the participants with a 10 ml syringe before the procedure. By attaching a 3-way tap to the injector from which the blood is drawn, blood is drawn into a second injector to ensure that the clotted blood is dispersed and homogenized. After the above-mentioned procedures, and after sufficient tissue samples were taken at the last stage of the biopsy procedure, control CT imaging, including the whole lung, was performed to evaluate complications. The presences of pneumothorax were noted. The prepared autologous blood patch was given through the coaxial needle (approximately 1 ml of autologous blood patch was applied for every 1 cm when the coaxial needle was withdrawn) and the tract formed by the biopsy needle in the parenchyma, pleura, and under the skin was closed with the participant's autologous blood. Thus, it was aimed at preventing pneumothorax or reducing its severity if it occurred. The tract formed by the given autologous blood patch into the parenchyma can be observed in most biopsies. The lesion and lung parenchyma features, pneumothorax and other complications of the participants included in the study were evaluated through biopsy planning and follow-up images in hospital medical record system. It is known that transthoracic lung biopsies performed with the coaxial technique increase the diagnostic accuracy. In addition, by obtaining more than one tissue piece with a single entry, more tissue pieces can be sampled for histopathological studies as well as molecular and genetic analysis, which has become increasingly important recently. As a result, investigators think that the use of this method will increase, as more tissue material can be obtained in percutaneous transthoracic lung biopsies performed with coaxial technique and computed tomography using the autologous blood patch method, while reducing the risk of pneumothorax, the most common complication, at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients who underwent percutaneous transthoracic tru cut biopsy
* Patients undergoing interventional procedures by radiologists with equal experience
* Patients who were able to obtain sufficient samples with the applied biopsy (technical success of percutaneous transthoracic biopsy)
* Patients whose medical records are fully accessible and whose data are reliable

Exclusion Criteria:

* Patients whose laboratory bleeding parameters are not suitable for the procedure (platelets<100000/mm3, INR>1.5)
* Pregnancy
* Patients with increased risk of pneumothorax due to other etiologies (bulla, blep, chronic obstructive pulmonary disease, cystic fibrosis)
* Patients receiving anticoagulant antiplatelet therapy
* Patients with persistent cough
* Patients with a history of recent lung travma, pneumothorax, hemoptysis or pulmonary hemorrhage
* Patients with severe psychiatric diseases such as psychosis or dementia that limit cooperation with the patient
* Patients with anatomic deformity (advanced scoliosis and kyphotic patients. Patients with pectus carinatum and pectus excavatum-like chest deformity)
* Patients for whom tru cut biopsy is absolutely and relative contraindicated (suspected hydatid cyst or known vascular lesions such as arteriovenous malformation, pulmonary varicose, severe obstructive pulmonary disease, coagulopathy, moderate to severe pulmonary hypertension, ventilator dependence, unilateral pneumectomy)
* Patients allergic to local anesthetic drug used for skin and subcutaneous tissue anesthesia
* Patients who do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study comprised 240 patients who received a transthoracic lung biopsy using the percutaneous coaxial technique at Trakya University Faculty of Medicine, Department of Radiology, Interventional Radiology unit, between January 1, 2015 and September 14, 2020.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Pneumothorax incidence | first 24 hours
  Development of pneumothorax after biopsy as a complication

SECONDARY OUTCOMES:
Chest tube placement incidence | Immediately after procedure
  Incidence of patients needing chest tube after biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Burak USLU, MD, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All patient data is stored in an institutionally encrypted medical system and cannot be shared openly.

REFERENCES:
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Result] Casal-Mourino A, Valdes L, Barros-Dios JM, Ruano-Ravina A. Lung cancer survival among never smokers. Cancer Lett. 2019 Jun 1;451:142-149. doi: 10.1016/j.canlet.2019.02.047. Epub 2019 Mar 6. PMID 30851418
- [Result] Marshall D, Laberge JM, Firetag B, Miller T, Kerlan RK. The changing face of percutaneous image-guided biopsy: molecular profiling and genomic analysis in current practice. J Vasc Interv Radiol. 2013 Aug;24(8):1094-103. doi: 10.1016/j.jvir.2013.04.027. Epub 2013 Jun 24. PMID 23806383
- [Result] Hiraki T, Mimura H, Gobara H, Shibamoto K, Inoue D, Matsui Y, Kanazawa S. Incidence of and risk factors for pneumothorax and chest tube placement after CT fluoroscopy-guided percutaneous lung biopsy: retrospective analysis of the procedures conducted over a 9-year period. AJR Am J Roentgenol. 2010 Mar;194(3):809-14. doi: 10.2214/AJR.09.3224. PMID 20173164
- [Result] Heerink WJ, de Bock GH, de Jonge GJ, Groen HJ, Vliegenthart R, Oudkerk M. Complication rates of CT-guided transthoracic lung biopsy: meta-analysis. Eur Radiol. 2017 Jan;27(1):138-148. doi: 10.1007/s00330-016-4357-8. Epub 2016 Apr 23. PMID 27108299